CLINICAL TRIAL: NCT07377656
Title: A Randomized, Observer-Blind, Placebo-Controlled, Proof-of-Concept Study to Assess the Safety, Tolerability and Immunogenicity of a Bivalent Human Papillomavirus (HPV) Vaccine in 9 and 15 Month Old Infants and Toddlers, 2-5 Year Old Children and an Open Label Single Dose Study in Young Unmarried Females Aged 15-20 Years in Ghana
Brief Title: Strengthening HPV Immunization Through EPI Leveraged Delivery
Acronym: SHIELD
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: International Vaccine Institute (Other)
Collaborators: Karolinska Institutet (Other); Noguchi Memorial Institute for Medical Research (Other); Dodowa Health Research Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IVI SHIELD 001
Record Dates: First submitted 2025-11-23; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: HPV Vaccine
Keywords: HPV; Proof of concept; Ghana; SHIELD; IVI; International Vaccine Institute; Karolinska Institutet; Dodowa Health Research Center
MeSH Terms: interventions — Papillomavirus Vaccines; Rubella Vaccine

STUDY DESIGN:
Intervention Model Description: This study follows an age de-escalation approach for the pediatric cohort. In the observer-blind arm, children aged 2-5 years will be enrolled first. Enrollment of the subsequent age groups will proceed only after DSMB review and approval at each stage. Following the first DSMB review and approval, enrollment of a limited number of participants aged 15 months will begin. After the next DSMB review and approval, recruitment will proceed for a subset of the 9-month-old age group while continuing enrollment in the 15-month cohort. A further DSMB review and approval will determine whether enrollment of the remaining 9-month-old participants may continue. Meanwhile, the open-label cohort of participants aged 15-20 years will begin enrollment concurrently with the 2-5-year-old group.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Arm AS (2-5 years old) (Experimental): HPV Vaccine
  Interventions: Biological: HPV vaccine
- Arm PS (2-5 years old) (Placebo Comparator): Placebo
  Interventions: Biological: Placebo
- Arm A15 (15 months old) (Experimental): HPV Vaccine
  Interventions: Biological: HPV vaccine; Biological: Measles and rubella Vaccine
- Arm P15 (15 months old) (Placebo Comparator): Placebo
  Interventions: Biological: Placebo; Biological: Measles and rubella Vaccine
- Arm A9 (9 months old) (Experimental): HPV + MR Vaccine
  Interventions: Biological: HPV vaccine; Biological: Measles and rubella Vaccine
- Arm P9 (9 months old) (Placebo Comparator): Placebo + MR Vaccine
  Interventions: Biological: Placebo; Biological: Measles and rubella Vaccine
- Arm E (15-20 years old) (Active Comparator): HPV Vaccine (Open Label)
  Interventions: Biological: HPV vaccine

INTERVENTIONS:
Biological: HPV vaccine — 0.5 mL HPV Vaccine Injection Intramuscular
  Arms: Arm A15 (15 months old); Arm A9 (9 months old); Arm AS (2-5 years old); Arm E (15-20 years old)
Biological: Placebo — 0.5 mL Placebo injection intramuscular
  Arms: Arm P15 (15 months old); Arm P9 (9 months old); Arm PS (2-5 years old)
Biological: Measles and rubella Vaccine — Measles and rubella Vaccine according to EPI
  Arms: Arm A15 (15 months old); Arm A9 (9 months old); Arm P15 (15 months old); Arm P9 (9 months old)

SUMMARY:
This is a randomized observer-blind placebo-controlled proof-of-concept study with the aim to assess the safety and tolerability, and the immunogenicity of a bivalent HPV vaccine administered in healthy infants and toddlers (9- and 15-month-olds) comparing them to an immune-bridging population of 15-20-year-old unmarried females in an open label study in Ghana at the Dodowa Health Research Center.

DETAILED DESCRIPTION:
Cervical cancer is a significant public health problem in Africa and a leading cause of cancer deaths in women. According to the WHO, Africa has the highest cervical cancer disease incidence and associated mortality in the world accounting for 19% of all global cases of cervical cancer and 23% of all cervical cancer related deaths. The high-risk Human Papillomavirus (HPV) Types16 and 18 are responsible for 70% of all global cervical cancers with a high prevalence of 22% in sub-Saharan Africa compared to a prevalence of 12%globally. The bivalent Cecolin HPV vaccine, manufactured by Innovax of China, has demonstrated >95% efficacy against HPV16/18 infections in women aged 18 to 26 years and some protection against HPV 31, 33 and 45. The hypothesis of this trial is that infants/toddlers vaccinated with the bivalent Cecolin will show similar safety, tolerability, and immunogenicity as compared to that observed in older age groups, 15 to 20year old, where efficacy has been established.

This trial is a proof-of-concept study to descriptively compare the safety, tolerability, and immunogenicity of HPV vaccination in a pediatric population. The aim is to demonstrate safety and tolerability, and that short-term immune responses in infants and toddlers are comparable to the responses in older girls and women between 15-20 years, an age group in whom efficacy has been shown. If the vaccines are shown to be safe, well tolerated, and sufficiently immunogenic in this pilot study, this would provide evidence to support larger statistically robust studies to test the safety, immunogenicity, longevity of immune response, and acceptability of including HPV vaccines in the routine EPI.

A total of one hundred and fifteen (N=115) eligible participants will be enrolled in the study with an age de-escalation approach for the pediatric cohort. First, the safety cohort of 15 children between the age of 2-5 years will be randomized in a 3:2 ratio to receive HPV (n=9) and placebo (n=6). To progress enrolment of toddlers aged 15 months, the DSMB will review safety data of the preceding safety cohort (2-5 years old) collected in the first week (until D7 visit) of follow-up according to pre-specified halting criteria. If halting criteria are not met, a further 15 toddlers (15 months) will be recruited similarly in a 3:2 ratio to receive HPV (n=9) and placebo (n=6). After the recruitment of the first 15 of 35 toddlers, there will be a second safety review by the DSMB. If halting criteria are not met, the remaining 20 participants of the 15-month-old cohort will continue recruitment. Following confirmation by the DSMB, 15 infants (9 months old) will be recruited similarly in a 3:2 ratio to receive HPV (n=9) and placebo (n=6). After the recruitment of the first 15 of 35 infants, there will be another safety review by the DSMB. If halting criteria are not met, the remaining 20 participants of the 9-month-old cohort will continue recruitment. The safety cohort and the toddlers will receive either a single dose of the HPV vaccine or placebo while the 9-month-old will either receive two doses of the HPV vaccine 6 months apart or the placebo. Adolescent girls and young women aged between 15 and 20 year olds will be recruited in open label study in parallel.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female individuals aged 9 months, 15 months, 2-5 years and unmarried females aged 15-20 years at the time of vaccination
* Participants aged 9 months, 15 months and 2-5 years who are up to date with their EPI vaccinations.
* Residing within the area of the study and planning to stay for the study duration.
* Participants that are HIV negative at screening (for the 9-15-month-olds a documented negative maternal ANC HIV screening).
* Unmarried females with a negative pregnancy test at screening practicing/willing to practice continuous effective contraception as recommended by the Ghana Health Services guidance in Ghana
* Able and willing to comply with all study requirements.
* Willingness to provide written informed consent before any trial procedure. Assent will be required for young female participants aged 15-17 years at vaccination in addition to their parent's/LAR's consent.

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Pregnancy, lactation, or intention to become pregnant during the vaccination phase through three months after the study vaccine dose
* Previous vaccination against HPV (Only for the 15-20-year-old efficacy cohort)
* Presence of malnutrition (weight-for-length z-score ≤-2SD median, per WHO published child growth standards)
* Planning to migrate out of the study areas before the end of the study follow-up
* Any underlying known condition or criteria, including acute or chronic clinically significant abnormality or infection that in the opinion of the investigator might compromise the wellbeing of the participant or interfere with the outcome of the study.
* Administration of immunoglobulins and/ or any blood products within the three months preceding the administration of the study vaccine.
* Known history of allergy or anaphylaxis to study vaccine components and/or excipients or other medications, or any other allergies deemed by the investigator to increase the risk of an adverse reaction.
* Any confirmed or suspected immunosuppressive or immunodeficient state, asplenia, recurrent severe infections and chronic use (more than 14 days) of immunosuppressant medication within 3 months prior to recruitment (topical steroids may be allowed).
* Any other finding that in the opinion of the investigators would increase the risk of an adverse outcome from participation in the trial or result in incomplete or poor-quality data.

Ages: 9 Months to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — For 15-20 years age group, only female participants will be enrolled. Other age groups (2-5 years old, 9 and 15 months old) both male and female participant will be enrolled.
Enrollment: 115 (Estimated)
Dates: Start 2026-01-16 (Estimated); Primary Completion 2028-02-29 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety and Reactogenicity of HPV Vaccination | 9 months post vaccination
  Occurrence of solicited and unsolicited adverse events following single-dose or two-dose HPV vaccination administered concomitantly with routine Expanded Programme on Immunization (EPI) vaccines, including Measles and Rubella (MR) vaccine, among infants aged 9 months, toddlers aged 15 months, and children aged 2-5 years. Results will be summarized as the number of participants experiencing adverse events
HPV16/18 VLP ELISA Antibody Titers | At 1, 7, 12, and 24 months post-HPV vaccination
  HPV16 and HPV18 antibody levels measured using Virus-Like Particle (VLP) Enzyme-Linked Immunosorbent Assay (ELISA) in serum samples collected from participants who received one or two doses of HPV vaccine. Antibody levels are expressed as ELISA antibody titers (IU/mL).
Geometric Mean Concentration of HPV16/18 Antibodies | At 1, 7, 12, and 24 months post-HPV vaccination
  Geometric mean concentration (GMC) of HPV16 and HPV18 antibodies measured using VLP ELISA in vaccinated participants, expressed as IU/mL.

SECONDARY OUTCOMES:
HPV16/18 Seroconversion Rate | 1 month and 7 months post HPV vaccination
  Seroconversion rate of HPV16 and HPV18 antibodies measured using VLP ELISA, defined as the proportion of participants who change from seronegative at baseline to seropositive after HPV vaccination. Results are expressed as a percentage of participants
HPV16/18 VLP ELISA Antibody Titers by Age and Sex | At 1, 7, 12, and 24 months post-HPV vaccination
  HPV16 and HPV18 antibody titers measured using VLP ELISA among male and female infants and toddlers aged 9 and 15 months and children aged 2-5 years following HPV vaccination, expressed as ELISA antibody titers (IU/mL).
Geometric Mean Concentration of HPV16/18 Antibodies by Age Group | At 1, 7, 12, and 24 months post-HPV vaccination
  Geometric mean concentration (GMC) of HPV16 and HPV18 antibodies measured using VLP ELISA among infants, toddlers, and children receiving HPV vaccination, expressed as IU/mL.
Measles and Rubella Seroconversion Rate | 1 month post MR vaccination
  Seroconversion rate of Measles and Rubella antibodies measured one month after MR vaccination among 9- and 15-month-old infants and toddlers who received MR vaccine with or without concomitant HPV vaccination. Results are expressed as a percentage of participants.

OTHER OUTCOMES:
HPV16/18 Neutralizing Antibody Titers (PBNA) | Baseline, 1, 7, 12, and 24 months post HPV vaccination
  Neutralizing antibody titers against HPV16 and HPV18 measured using a pseudovirion-based neutralization assay (PBNA) in participants who received one or two doses of HPV vaccine. Results are expressed as neutralizing antibody titers.
Geometric Mean Concentration of HPV16/18 Neutralizing Antibodies | Baseline, 1, 7, 12, and 24 months post HPV vaccination
  Geometric mean concentration of neutralizing antibodies against HPV16 and HPV18 measured using PBNA, expressed as geometric mean neutralizing antibody titers.
Acceptability of HPV Vaccination in Infants and Toddlers | Up to 7 months post vaccination
  Acceptability of HPV vaccination in infants and toddlers as reported by parents or caregivers and healthcare workers using structured questionnaires, summarized using questionnaire scores

CONTACTS AND LOCATIONS:
Overall Officials: Julia Lynch, MD, Study Director — International Vaccine Institute; George Armah, Prof. PhD, Principal Investigator — Noguchi Memorial Institute for Medical Research
Locations (1):
- Dodowa Health Research Center, Accra, Ghana

IPD SHARING:
Plan to Share IPD: No